CLINICAL TRIAL: NCT07269236
Title: Prospective Real-World Study of a Multimodal Artificial Intelligence Model Across Disease Types
Brief Title: Prospective Real-World Study of Multimodal AI
Status: Enrolling by invitation | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-602
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Pancancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples Without DNA: Samples retained, with no potential for DNA extraction from any retained samples (e.g., fixed tissue, plasma)

GROUPS / COHORTS (3):
- ZSCPH validation dataset: Approximately 1,000 prospective patients across various disease types will have digitized scanned images, imaging information, and clinicopathological data provided, collected from Zhongshan People's Hospital (Zhongshan, Guangdong, China) between October 2025 and September 2030.
- NFHSMU validation dataset: We conducted a prospective validation study to compare the diagnostic performance among pathologists, our multimodal artificial intelligence model . This study was initiated on October 1, 2025 at Nanfang Hospital, Southern Medical University (NFHSMU).
- Randomized controlled trial: We conducted a prospective randomized controlled trial to compare the diagnostic performance among pathologists, the multimodal artificial intelligence model, and pathologist-with-model-assisted diagnosis at Nanfang Hospital of Southern Medical University (NFHSMU).The trial commenced data collection on October 1, 2025 to establish the NFHSMU randomized controlled trial dataset. Following quality control, the slides were randomly allocated (1:1:1 ratio) into three groups:Model-only group/Pathologist-only group/Model-assisted pathologist group.

SUMMARY:
This project proposes to collect prospective multimodal data-such as pathology, imaging, and clinical information-and to perform integrative analyses. AI technologies can offer novel solutions for disease classification, tumor grading, histological subtyping, molecular subtyping, selection of chemotherapy regimens, risk stratification, treatment response prediction, report generation, and intelligent question-answering. This research provides important support for precision medicine and individualized treatment and has significant theoretical and practical implications. Conducting a prospective randomized controlled study better aligns with clinical application requirements and can accelerate the comprehensive deployment of AI systems.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Patients with available digitized pathology slides, radiological imaging, and corresponding clinical data.

Exclusion Criteria:

1.Patients with missing data or specimens not meeting quality control requirements for analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria comprised patients with definitive pathological diagnoses. All cases were prospectively collected from Nanfang Hospital, Southern Medical University (NFHSMU) .
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Area under ROC curve (AUC) | Diagnostic evaluation will be performed within 1 week when the WSIs or CT are obtained
  Area under the curve

SECONDARY OUTCOMES:
Specificity | Diagnostic evaluation will be performed within 1 week when the WSIs or CT are obtained
  The true negative rate (TNR) of the diagnostic platform, which is the ratio between the number of negative individuals correctly categorized by platform and the total number of actual negative individuals (%).
Sensitivity | Diagnostic evaluation will be performed within 1 week when the WSIs or CT are obtained
  The true positive rate (TPR) of the diagnostic platform, which is the ratio between the number of positive individuals correctly categorized by platform and the total number of actual positive individuals (%).

CONTACTS AND LOCATIONS:
Overall Officials: Li Liang, Study Director — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong

IPD SHARING:
Plan to Share IPD: No
Requests for the data collected and analyzed in this study will be considered if the application is in line with public benefits and the applicant is willing to sign a data access agreement. Contact can be through the corresponding author.